CLINICAL TRIAL: NCT01299038
Title: A Multi-dose Phase II Trial of Rosuvastatin to Lower Circulating Tissue Factor Bearing Microparticles in Metastatic Breast Cancer
Brief Title: Rosuvastatin to Lower Circulating Tissue Factor Bearing Microparticles in Metastatic Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Beth Israel Deaconess Medical Center (Other)
Collaborators: Dana-Farber Cancer Institute (Other); Massachusetts General Hospital (Other); National Institutes of Health (NIH) (NIH)
Responsible Party: Principal Investigator, Jeffrey Zwicker, MD, Assistant Professor, Harvard Medical School, Dana-Farber Cancer Institute
Organization: Dana-Farber Cancer Institute (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 10-287
Record Dates: First submitted 2011-02-16; First posted 2011-02-18 (Estimated); Results first posted 2020-02-05 (Actual); Last update posted 2020-02-05 (Actual); Status verified 2020-01

CONDITIONS: Breast Cancer
Keywords: Crestor; TFBP; rosuvastatin
MeSH Terms: conditions — Breast Neoplasms | interventions — Rosuvastatin Calcium

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group 1 (Active Comparator): Rosuvastatin 20mg taken orally once a day for 4 weeks
  Interventions: Drug: rosuvastatin
- Group 2 (Active Comparator): Rosuvastatin 40mg taken orally once a day for 4 weeks
  Interventions: Drug: rosuvastatin

INTERVENTIONS:
Drug: rosuvastatin — Taken orally once a day for 4 weeks
  Other Names: Crestor

SUMMARY:
Research studies have shown a strong association between cancer and blood clots in the veins (also known as deep vein thrombosis). These blood clots can flow to the lungs (pulmonary embolism) which in severe cases may be life threatening. Studies have demonstrated that increases in microparticles may contribute to the development of deep vein thrombosis in cancer patients. The purpose of this research study is to see if rosuvastatin lowers the number of tissue factor bearing microparticles in the blood (TFMP). TFMP are small particles that are generated from different types of blood cells in the body. In people who have cancer, TFMP are thought to be generated from cancer cells and may represent a risk factor for deep vein thrombosis.

DETAILED DESCRIPTION:
* Since no one knows which of the study options are best, participants will be "randomized" into the following study groups: Group 1 (regular dose of rosuvastatin) or Group 2 (higher dose of rosuvastatin).
* Participants will take 1 pill of rosuvastatin every day for 4 weeks. Each 4 week period is called a cycle.
* Participants will have a physical exam at baseline, on day 1 of starting rosuvastatin, and 2 month visits. Laboratory tests will be taken at baseline, on day 1 of starting rosuvastatin, 6 weeks and 2 months.

ELIGIBILITY:
Inclusion Criteria:

* Metastatic adenocarcinoma of the breast (Stage IV)
* Actively receiving endocrine therapy for at least 6 weeks (with or without HER2 therapy)
* Minimum age 18 years
* ECOG Performance status of 0, 1 or 2
* Normal organ and marrow function as defined in the protocol

Exclusion Criteria:

* Participants may not be receiving any other study agents
* Actively receiving chemotherapy (exclusive of hormonal or HER2 therapy ) within last 5 weeks
* Any statin therapy within the last 3 weeks
* Asian decent (including Filipino, Chinese, Japanese, Korean, Vietnamese or Asian-Indian origin)
* Concomitant use of the following drugs: cyclosporine, fibrates, niacin, gemfibrozil, ketaconazole, spironolactone, cimetidine, warfarin, erythromycin, or protease inhibitors
* Conditions predisposing to renal failure secondary to rhabdomyolysis
* Recent history of heavy alcohol use as judged by the treating physician
* Known to be pregnant (testing not required) or nursing
* History of rhabdomyolysis on statin therapy
* Known history of Hepatitis C or active hepatitis B infection (baseline testing not required)
* Uncontrolled intercurrent illness including, but not limited to ongoing or active infection, hepatitis, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2010-10 (Actual); Primary Completion 2013-11 (Actual); Study Completion 2013-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey I. Zwicker, MD, Principal Investigator — Beth Israel Deaconess Medical Center
Locations (2):
- United States (2):
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts

RESULTS

PARTICIPANT FLOW:
Groups:
- Rosuvastatin 20: Rosuvastatin 20mg taken orally once a day for 4 weeks
- Rosuvastatin 40: Rosuvastatin 40mg taken orally once a day for 4 weeks
Period: Overall Study
Arm/Group | Rosuvastatin 20 | Rosuvastatin 40
Started | 10 (Consented) | 10 (Consented)
Completed | 9 (Evaluable) | 10 (Evaluable)
Not Completed | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Population: The analysis of dataset is comprised of all evaluable patients.
Groups:
- Rosuvastatin 20mg: Rosuvastatin 20mg taken orally once a day for 4 weeks
  rosuvastatin: Taken orally once a day for 4 weeks
- Rosuvastatin 40mg: Rosuvastatin 40mg taken orally once a day for 4 weeks
  rosuvastatin: Taken orally once a day for 4 weeks
- Total: Total of all reporting groups
Arm/Group | Rosuvastatin 20mg | Rosuvastatin 40mg | Total
Number analyzed (Participants) | 9 | 10 | 19
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 8 | 7 | 15
  >=65 years | 1 | 3 | 4
Sex/Gender, Customized [Number; unit: participants]
  Female | 9 | 10 | 19
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 9 | 10 | 19
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Mean Change of Tissue Factor Bearing Microparticles
Description: Comparison of plasma microparticle concentration between baseline and week 4
Time Frame: 4 weeks
Measure: Mean (Standard Deviation); unit: microparticles per microliter
Arm/Group | Rosuvastatin 20mg | Rosuvastatin 40mg
Number analyzed (Participants) | 8 | 7
microparticles per microliter | 102 (586) | -618 (624)

ADVERSE EVENTS:
Time Frame: Assessed during the 4 weeks therapy
Arm/Group | Rosuvastatin 20mg | Rosuvastatin 40mg
Serious Adverse Events (participants affected / at risk) | 0/9 | 0/10
Other Adverse Events (participants affected / at risk) | 9/9 | 9/10
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Rosuvastatin 20mg (N=9) | Rosuvastatin 40mg (N=10)
Pain (General disorders) | 0 | 3 — Joint and muscle pain
Edema limbs (General disorders) | 1 | 1
Chills (General disorders) | 1 | 0
Hypercalcemia (Metabolism and nutrition disorders) | 1 | 0
Hypertension (Vascular disorders) | 2 | 0
Hyperuricemia (Metabolism and nutrition disorders) | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 1
Headache (Nervous system disorders) | 2 | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 2
General disorders and administration site conditions - Other, specify (General disorders) | 0 | 1 — Right leg numbness
Leukocytosis (Blood and lymphatic system disorders) | 0 | 1
Alanine aminotransferase increased (Investigations) | 0 | 1
Aspartate aminotransferase increased (Investigations) | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 4
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 1 | 0
Platelet count decreased (Investigations) | 0 | 1
Hot flashes (Vascular disorders) | 1 | 3
Gastric ulcer (Gastrointestinal disorders) | 0 | 1
Upper respiratory infection (Infections and infestations) | 0 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 1
Arthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1
Paresthesia (Nervous system disorders) | 1 | 0
Hypermagnesemia (Metabolism and nutrition disorders) | 1 | 0
Iron overload (Metabolism and nutrition disorders) | 1 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 1 | 0
Hyperthyroidism (Endocrine disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 1 | 1
Gastroesophageal reflux disease (Gastrointestinal disorders) | 1 | 1
Thrombotic thrombocytopenic purpura (Blood and lymphatic system disorders) | 1 | 0
Encephalopathy (Nervous system disorders) | 1 | 0
Hypokalemia (Metabolism and nutrition disorders) | 0 | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Palpitations (Cardiac disorders) | 0 | 1
Sinus tachycardia (Cardiac disorders) | 1 | 0
Fatigue (General disorders) | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dizziness (Nervous system disorders) | 0 | 1
Ascites (Gastrointestinal disorders) | 0 | 1
Peripheral sensory neuropathy (Nervous system disorders) | 1 | 0
Nightmares (General disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No